CLINICAL TRIAL: NCT07180199
Title: Evaluation of the Results of Surgical Correction of V Pattern Intermittent Exotropia Without Inferior Oblique Muscle Overaction
Brief Title: Surgical Correction of V Pattern Intermittent Exotropia Without Inferior Oblique Muscle Overaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sarah Abdelrahman Abdelwahab Oun, Resident at Ophthalmology Department, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264MS244/7/23
Record Dates: First submitted 2025-09-11; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Surgical Correction; V Pattern; Intermittent Exotropia; Inferior Oblique Muscle; Overaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilateral Lateral Rectus Recession (BLR Recession) (Experimental): Participants underwent bilateral lateral rectus recession procedure alone for correction of large-angle exotropia.
  Interventions: Procedure: Bilateral Lateral Rectus Recession (BLR Recession)
- Bilateral Lateral Rectus Recession with Upward Transposition (Experimental): Participants underwent bilateral lateral rectus recession combined with upward transposition of the muscle insertion to enhance alignment in cases of large-angle exotropia.
  Interventions: Procedure: Bilateral Lateral Rectus Recession with Upward Transposition

INTERVENTIONS:
Procedure: Bilateral Lateral Rectus Recession (BLR Recession) — This procedure involved recession of both lateral rectus muscles to reduce large-angle exotropia.
  Arms: Bilateral Lateral Rectus Recession (BLR Recession)
Procedure: Bilateral Lateral Rectus Recession with Upward Transposition — This procedure involved bilateral lateral rectus recession combined with upward transposition of the insertion to enhance ocular alignment in patients with large-angle exotropia.
  Arms: Bilateral Lateral Rectus Recession with Upward Transposition

SUMMARY:
Evaluation of the results of surgical correction of V pattern intermittent exotropia without inferior oblique muscle overaction by either performing bilateral lateral rectus recession (BLR) alone or performing bilateral lateral rectus recession asssosiated with upward transposition of lateral rectus muscle insertion

DETAILED DESCRIPTION:
Intermittent exotropia (IXT) is the most common type of strabismus which is a disorder of binocular eye movement control in which one eye intermittently moves outwards.Intermittent exotropia may be associated with difference in the horizontal deviation from the primary position to the upward or downward gaze giving A or V pattern In V-pattern intermittent exotropia (XT), there is an increase in the horizontal deviation as the eyes move from downgaze to upgaze.

Non-surgical treatment includes correction of refractive error, orthoptics, overcorrecting minus lenses and prismotherapy. Surgical options includes unilateral medial rectus muscle resection combined with a lateral rectus muscle recession or bilateral lateral rectus recession as in basic type IXT OR bilateral lateral rectus muscle recession as in divergent excess type OR bilateral medial rectus muscle resection as in convergence insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Patients with V pattern intermittent exotropia (XT increasing by >10Δ in upgaze compared with Downgaze).
* No or minimal inferior oblique overaction on both sides (+1)
* Minimum follow-up period of 6 months after surgical correction of strabismus

Exclusion Criteria:

* Structural eye pathology.
* Significant neurodevelopmental delay.
* ntermittent exotropia without V pattern.
* Superior oblique under action.
* Duane syndrome.
* Less than 6 months follow up.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Angle of Ocular Deviation | 6 months postoperatively
  The degree of ocular misalignment was measured using prism cover test at near and distance fixation. Successful outcome was defined as residual deviation ≤10 prism diopters.

SECONDARY OUTCOMES:
Postoperative Complications | 6 months postoperatively
  Complications such as overcorrection, undercorrection, or limitation of ocular motility were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia Governorate, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author